CLINICAL TRIAL: NCT03660319
Title: The Effect of EMT on Anxiety Levels and Perception of Waiting Time in the Radiation Oncology Waiting Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1190
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cancer
Keywords: music therapy; EMT; environmental music therapy; radiation oncology; anxiety; waiting room
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants randomized into two groups: Music Therapy Intervention (Environmental Music Therapy) and Control arm with no Music Therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Environmental Music Therapy (Experimental): Music Therapy Intervention (EMT)
  Interventions: Other: Environmental Music Therapy
- Control (No Intervention): Control - No Environmental Music Therapy. Does not experience Environmental Music Therapy during wait time in radiation oncology waiting room.

INTERVENTIONS:
Other: Environmental Music Therapy — Experiencing Environmental Music Therapy during wait time in radiation oncology waiting room.
  Other Names: Music Therapy Intervention
  Arms: Environmental Music Therapy

SUMMARY:
This study will be investigating the effects of environmental music therapy (EMT) on patient and caregiver anxiety levels and perceptions of waiting time for patients undergoing radiation therapy. Environmental music therapy is live music offered by a music therapist with the intention of modifying patients' and caregivers' perception of the environment itself and in so doing provide an experience of enhanced comfort and relaxation. One hundred and sixty patients and their caregivers, when present, who are diagnosed with Cancer, including head & neck, breast, prostate, lymphoma, gastro-intestinal, and skin cancers, as well as other cancers will be identified and referred by Mount Sinai Downtown radiation oncology attending doctors prior to their arrival in the waiting room of the Radiation Oncology Suite. All Cancer subjects will be considered regardless of gender or racial/ethnic background, and health status with the exception of those less than 18 years of age. Only patients who are fluent in English will be eligible to enroll in the study. Patients will randomly be assigned to the control or environmental music group. The patients in the control group will be able to receive music therapy during radiation therapy, even though they will not have music therapy during their waiting room time, as is the focus of this study.

DETAILED DESCRIPTION:
Objectives:

Will EMT affectively reduce state anxiety and time distortion in patients receiving radiation therapy for cancer and in their personal caregivers during their time in the radiation oncology department waiting room? The purpose of this study is to (a) rate the patients level of anxiety and discomfort prior to radiation therapy as experienced in the waiting area, (b) determine if the following music psychotherapy protocol moderates baseline anxiety related to their treatment experience and (c) evaluate how an environmental music therapy protocol affects the subjects' perception of the amount of they have waited before treatment measured against the actual amount of time they have waited.

Hypothesis:

EMT will reduce state anxiety and time distortion for cancer patients and their personal caregivers in the radiation oncology waiting room.

The current study will focus on effects of music therapy on 160 patients and their caregivers, who are randomly assigned to two groups. All patients with cancer who receive radiation and who are waiting for radiation therapy in the waiting room are eligible, with the exception of those patients who are not fluent in English. Enrolled participants will complete the abridged State Trait Anxiety Inventory and the Wong-Baker faces scale pre and post EMT or no EMT. The music therapist will provide prescribed live patient-preferred music in conjunction with the patients' culture, past medical history, past trauma, and assessment of psychological stressors to be observed and expressed prior to radiation, as they wait in the waiting room. The live music used will provide an anchor and suggest inter-relationship possibilities amongst patients and their caregivers during the EMT sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Receiving treatment for cancer in the radiation oncology department
* Personal caregivers of patients receiving treatment for care in the radiation oncology department

Exclusion Criteria:

* Adults who are not fluent in English
* Adults unable to consent
* Individuals who are not yet adults (e.g. infants, children, teenagers)
* Wards of the State (e.g. foster children)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Scale | Day 1
  Anxiety measured by Wong-Baker Faces Scale during their waiting which has 6 faces with the first face scored 0 (no anxiety) to the last face scored 10 (high anxiety), total scale from 0-10, higher score indicating more anxiety
Short-Form STAI | Day 1
  Anxiety measured by Short-Form STAI during their waiting. Short-Form STAI is a 6-item instrument. To calculate the total STAI score (range 20 - 80):
  * reverse scoring of the positive items (calm, relaxed, content) so 1=4, 2=3, 3=2 and 4=1;
  * sum all six scores;
  * multiply total score by 20/6; with higher score indicating more anxiety

SECONDARY OUTCOMES:
Perceived Waiting Time | Day 1
  Perception of waiting time questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rossetti, MMT, Study Chair — Icahn School of Medicine at Mount Sinai; Joanne Loewy, DA, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Downtown Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No